CLINICAL TRIAL: NCT07202299
Title: Randomized Controlled Trial of Two Protocols for Weaning From High Frequency Oscillatory Ventilation in Preterm Neonates With Respiratory Distress Syndrome
Brief Title: Open-label Randomized Controlled Trial of Two Protocols for Weaning From High Frequency Oscillatory Ventilation in Preterm Neonates With Respiratory Distress Syndrome Admitted in the NICU of Mansoura University Children Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Yasmina Elsaied Hassan Keshta, assistant lecturer of pediatrics, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD.25.05.1000
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Distress Syndrome (Neonatal)
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (intervention group) (Experimental): Group I (Intervention group): Fifty five preterm infants with direct weaning from HFOV (high frequency oscillatory ventilation) to CPAP (continuous positive airway pressure).
  Interventions: Other: HFOV weaning protocol 1
- Group II (Control group) (Active Comparator): Group II (Control group): Fifty five preterm infants with weaning from HFOV (high frequency oscillatory ventilation) to conventional mechanical ventilation (CMV) then to CPAP (continuous positive airway pressure) .
  Interventions: Other: HFOV weaning protocol 2

INTERVENTIONS:
Other: HFOV weaning protocol 1 — weaning preterm neonates with RDS from HFOV directly to CPAP
  Arms: Group 1 (intervention group)
Other: HFOV weaning protocol 2 — weaning of preterm neonates with RDS to CMV then to CPAP
  Arms: Group II (Control group)

SUMMARY:
Our study is a randomized controlled trial that compares two weaning protocols of preterm infants with respiratory distress syndrome who are ventilated on high frequency oscillatory ventilation in order to establish the best weaning strategy with the least complications possible for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with RDS whose gestational age is 34 weeks or less who required HFOV for more than 24 hours duration due to failure of non- invasive respiratory support due to any of the following:

  1. Severe hypercapnea PaCO2 > 60 mmHg associated with pH < 7.25.
  2. Hypoxemia PaO2 < 50 mmHg, with FiO2 > 40%.
  3. Frequent apneas: 6 or more episodes of apnea requiring mild or moderate stimulation within 6-hour period or one apneic episode requiring bag and mask positive pressure ventilation.

Exclusion Criteria:

Preterm infants with any of the following :

1. Major congenital malformations or chromosomal aberrations.
2. Inborn errors of metabolism.
3. Severe intraventricular hemorrhage (IVH) grade III or IV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
comparing weaning failure rate between 2 groups | 72 hours after weaning
  Failure of weaning will be considered if the infant develops respiratory distress again requiring re-intubation within 72 hours after extubation due to any of the following:
  1. Severe hypercapnia (PaCO2 > 60 mmHg) .
  2. Hypoxemia ( PaO2 < 50 mm Hg).
  3. Frequent apnea (6 apnea episodes within 6-hour period or 1 apneic episode requiring bag and mask positive pressure ventilation).
     Or escalation of respiratory support as following:
  4. Titration of CPAP level out of the assigned range (CPAP pressure > 8 cmH2O).
  5. Escalation to an alternate mode of non-invasive respiratoy support such as non-invasive positive pressure ventilation (NIPPV).

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided